CLINICAL TRIAL: NCT06681818
Title: Postoperative Heme Oxygenase Induction and Carbon Monoxide Production as a Novel Method to Assess Hepatic Regeneration and Predict Hepatic Related Morbidity After Partial Hepatectomy
Brief Title: Novel Method to Assess Hepatic Regeneration and Predict Hepatic Related Morbidity After Partial Hepatectomy
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Englewood Hospital and Medical Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: E-24-982
Record Dates: First submitted 2024-11-06; First posted 2024-11-08 (Actual); Last update posted 2025-07-23 (Actual); Status verified 2024-11

CONDITIONS: Liver Cancer Adult; Liver Regeneration
Keywords: hepatectomy
MeSH Terms: conditions — Carcinoma, Hepatocellular

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- all participants (Experimental): all participants will provide breath samples to detect carbon monoxide levels
  Interventions: Other: carbon monoxide measurement via smokerlyzer

INTERVENTIONS:
Other: carbon monoxide measurement via smokerlyzer — participants in this study will provide breath samples for carbon monoxide measurements pre and post liver resection

SUMMARY:
the investigators will pursue two specific aims: (1) to monitor the extent of heme oxygenase induction (by measuring endogenous CO production) in relationship to the extent of hepatic resection (2) to assess the production of CO in patients following liver resection and correlate these findings to the rate of liver regeneration and liver function.

ELIGIBILITY:
Inclusion Criteria:

* Patient plans to have partial liver resection for primary liver pathology or metastatic disease
* Patient is able to comprehend and willing to sign the written consent form

Exclusion Criteria:

* Patients < 18 years
* Patients identified as members of a vulnerable population, except women of child bearing potential with negative pregnancy test

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 125 (Estimated)
Dates: Start 2025-11-21 (Estimated); Primary Completion 2039-01-01 (Estimated); Study Completion 2039-01-01 (Estimated)

PRIMARY OUTCOMES:
correlation of carbon monoxide levels in exhaled breath with quantity and quality of liver regeneration | measurements will be taken pre, then 4 hours and 24 hours post resection
  patients will be asked to donate exhaled breath into a smokerlyzer device

SECONDARY OUTCOMES:
level of carbon monoxide in exhaled air of patients | measurements will be taken pre, then 4 hours and 24 hours post resection
  patients will be asked to donate exhaled breath into a smokerlyzer device
quantity of liver regeneration, liver volume (ml) | one and three months after resection
  CT liver volumetric studies
quality of hepatic regeneration, normalized liver function | one and three months post resection
  serum protein, albumin, AST and ALT, alkaline phosphatase, and bilirubin level

CONTACTS AND LOCATIONS:
Overall Officials: Cherif Boutros, MD, Principal Investigator — Englewood Hospital
Locations (1):
- Englewood Hospital, Englewood, New Jersey, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Related Info — https://www.englewoodhealth.org/